CLINICAL TRIAL: NCT05950581
Title: Treatment Skeletal Class II Malocclusion With Modified Twin-Block Appliance With Clear Plates VS Traditional Twin Block
Brief Title: Treatment of Skeletal Class II Malocclusion With Modified Twin-Block Appliance With Clear Plates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hama University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hama University -Orthdontic.
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- : Modified Twin-Block Appliance with Clear Plates. (Experimental): Clear plates technique A group of patients in which participants will be undergo to clear plates treatment will be applied to the upper and lower arch 17 hours daily Experimental : Modified Twin-Block Appliance with Clear Plates.
  Interventions: Device: Modified Twin-Block Appliance with Clear Plates.
- Traditional Twin-Block appliance (Experimental): Traditional Twin-Block appliance A group of patients in which participants will undergo to the Traditional Twin-Block appliance Treatment, appliances will be applied to the upper and lower arch 17 hours daily
  Interventions: Device: Traditional Twin-Block appliance

INTERVENTIONS:
Device: Modified Twin-Block Appliance with Clear Plates. — Clear plates technique A group of patients in which participants will be undergo to clear plates treatment will be applied to the upper and lower arch 17 hours daily
  Arms: : Modified Twin-Block Appliance with Clear Plates.
Device: Traditional Twin-Block appliance — Traditional Twin-Block appliance A group of patients in which participants will undergo to the Traditional Twin-Block appliance Treatment, appliances will be applied to the upper and lower arch 17 hours daily
  Arms: Traditional Twin-Block appliance

SUMMARY:
Patients with skeletal class II malocclusion who have a retracted lower jaw will be treated in this study. The efficacy of clear Plates in the treatment of Skeletal Class II Malocclusion will be assessed. The skeletal, dental and soft tissues changes resulted by this intervention will be studied and compared with the results of Traditional treatment with fixed appliances.

DETAILED DESCRIPTION:
There are two group:

1. a group of patients in which participants will be undergo to Modified Twin-Block Appliance with Clear Plates.
2. a group of patients in which participants will be undergo to the traditional Twin-Block Appliance.

phase Intervention/treatment Condition or disease

Not applicable Other:

Modified Twin-Block Appliance with Clear Plates.

Other:

Traditional Twin-Block Appliance. Skeletal class II Malocclusion

ELIGIBILITY:
Inclusion Criteria:

* - Patients with mixed dentition at age 10.5-13 years.
* The patient has Skeletal class II malocclusion caused by mandibular retraction ANB > 5, 8 mm >O.J> 5 mm, SNB<78, angle (NSAr) ≥ ° 125 and normal placement of the upper jaw.
* The patient is willing to accept treatment with a removable device.
* No previous orthodontic treatment
* the growth model is within the normal or horizontal maxillary opening angle of 30 >MM or angle of 400 > Björk
* patients do not have an upper alveolar dental protrusion.

Exclusion Criteria:

* -Patients with periodontal disease.
* patients with a neuromuscular disorder.
* patients of class I or III of malocclusion.
* Patients with temporomandibular joint disorder.
* Patients with Skeletal open bite.
* Patients with poor oral and gingival health
* the presence of a unilateral or bilateral posterior crossbite.
* patients who have upper jaw stenosis and need to be prepared by expansion before functional treatment.
* any patient who does not meet one or more of the Inclusion criteria will be removed from the study.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in the SNA angle[ | : T0:1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6-9 months in the exp. Group and control group)
  This angle the represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in the SNB angle [ | : T0:1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6-9 months in the exp. Group and control group)
  This angle the represents the position of the lower jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in the mandibular length | T0: 1day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6-9 months in the exp. Group and control group)
  Amount of distance measured from the Co point to Gn point in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in overjet | T0: 1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6-9 months in the exp. Group and control group)
  Represents The distance between the most anterior point on the lower incisor to the most anterior point on the upper incisor in the cephalometric analysis.
change in the vertical position of incisors | : T0: 1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 6-9 months in the exp. Group and control group)
  The vertical distance from the edge of the lower incisor to the mandibular plane.

CONTACTS AND LOCATIONS:
Overall Officials: Rabab Alsabbagh,, DDS MSc PhD, Study Director — Professor of Orthodontics, University of Hama Dental School, Hama, Syria.; ANAS FAKHOURI, Principal Investigator — Student in Orthodontics, University of Hama Dental School, Hama.
Locations (1):
- Hama University, Hama, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buschang PH, Stroud J, Alexander RG. Differences in dental arch morphology among adult females with untreated Class I and Class II malocclusion. Eur J Orthod. 1994 Feb;16(1):47-52. doi: 10.1093/ejo/16.1.47. PMID 8181550
- [Background] Clark WJ. The twin block technique. A functional orthopedic appliance system. Am J Orthod Dentofacial Orthop. 1988 Jan;93(1):1-18. doi: 10.1016/0889-5406(88)90188-6. No abstract available. PMID 3422118
- [Background] Cozza P, Baccetti T, Franchi L, De Toffol L, McNamara JA Jr. Mandibular changes produced by functional appliances in Class II malocclusion: a systematic review. Am J Orthod Dentofacial Orthop. 2006 May;129(5):599.e1-12; discussion e1-6. doi: 10.1016/j.ajodo.2005.11.010. PMID 16679196
- [Background] de Lira Ade L, de Moura WL, Artese F, Bittencourt MA, Nojima LI. Surgical prediction of skeletal and soft tissue changes in treatment of Class II. J Craniomaxillofac Surg. 2013 Apr;41(3):198-203. doi: 10.1016/j.jcms.2012.07.009. Epub 2012 Nov 30. PMID 23201327
- [Background] Fritz JD, Utz AL, Hale NM, Wu L, Powers AC, Verdoorn TA, Robertson D. Gene-based neurotransmitter modulation in cerebellar granule neurons. J Neurochem. 1997 Jan;68(1):204-12. doi: 10.1046/j.1471-4159.1997.68010204.x. PMID 8978727
- [Background] Trenouth MJ. Cephalometric evaluation of the Twin-block appliance in the treatment of Class II Division 1 malocclusion with matched normative growth data. Am J Orthod Dentofacial Orthop. 2000 Jan;117(1):54-9. doi: 10.1016/s0889-5406(00)70248-4. PMID 10629520
- [Background] Tulloch JF, Medland W, Tuncay OC. Methods used to evaluate growth modification in Class II malocclusion. Am J Orthod Dentofacial Orthop. 1990 Oct;98(4):340-7. doi: 10.1016/S0889-5406(05)81491-X. PMID 2220695